CLINICAL TRIAL: NCT06460493
Title: A Study Assessing the Effect of Ensifentrine on CAT™ Scores Over 12 Weeks in Subjects With Moderate to Severe COPD
Brief Title: Effect of Ensifentrine Treatment on CAT Score
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Verona Pharma plc (Industry)
Collaborators: Midwest Chest Consultants (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RPL554-CO-303
Record Dates: First submitted 2024-06-10; First posted 2024-06-14 (Actual); Results first posted 2025-04-18 (Actual); Last update posted 2025-04-18 (Actual); Status verified 2025-03

CONDITIONS: COPD
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — ensifentrine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Ensifentrine (Experimental): Inhaled ensifentrine twice daily for 12 weeks via standard jet nebulizer in addition to standard dual (LAMA/LABA) or triple (LAMA/LABA/ICS) COPD therapy.
  Interventions: Drug: Ensifentrine 3 mg twice daily

INTERVENTIONS:
Drug: Ensifentrine 3 mg twice daily — All subjects will receive ensifentrine.
  Other Names: RPL554

SUMMARY:
The purpose of this open-label, single center trial is to assess the effect of twice daily nebulized ensifentrine (3 mg) on COPD symptoms measured by the COPD Assessment Test (CAT™) scores over 12 weeks in subjects with symptomatic, moderate to severe COPD, taking maintenance LAMA/LABA or LAMA/LABA/ICS therapy. Subjects will continue the maintenance treatment during study participation.

ELIGIBILITY:
Inclusion Criteria:

* Capable of giving informed consent.
* Current or former cigarette smokers with a history of cigarette smoking ≥ 10 pack years.
* Established clinical history of moderate to severe COPD.
* Pre- and post-albuterol FEV1/FVC ratio of < 0.70.
* Post-albuterol FEV1 ≥ 30 % and ≤ 75% of predicted normal.
* ≥2 on the modified Medical Research Council (mMRC) Dyspnea Scale.
* ≥10 on the COPD Assessment Test™.
* Taking stable dual (LAMA+LABA) or triple (LAMA+LABA+ICS) maintenance therapy for at least 8 weeks.
* Capable of using a standard jet nebulizer and performed spirometry assessment.

Exclusion Criteria:

1. Hospitalizations for COPD (or COPD exacerbation), pneumonia, or other serious infection or treatment with oral or parenteral (oral, intravenous, or intramuscular) glucocorticoids within the past 12 weeks.
2. Lower respiratory tract infection within the past 6 weeks or an active infection.
3. History of life-threatening COPD, including Intensive Care Unit admission and/or requiring intubation within 1-year.
4. Major surgery (requiring general anesthesia) within the past 6 weeks, lack of full recovery from surgery, or planned surgery through the end of the study.
5. Concomitant clinically significant pulmonary disease other than COPD (e.g., asthma, tuberculosis, lung cancer, bronchiectasis, sarcoidosis, lung fibrosis, interstitial lung diseases, sleep apnea (unless controlled with stable continuous positive airway pressure [CPAP] use), known alpha-1 antitrypsin deficiency, core pulmonale or other non-specific pulmonary disease).
6. Severe comorbidities including unstable cardiac, (e.g., myocardial infarction within 1 year prior to screening, unstable angina within 6 months, or unstable or life-threatening arrhythmia requiring intervention within 3 months) or any other clinically significant medical conditions including uncontrolled diseases (e.g., endocrine, neurological, hepatic, gastrointestinal, renal, hematological, urological, immunological, psychiatric or ophthalmic diseases) that would, in the opinion of the Investigator, preclude the subject from safely completing the required tests or the study, or is likely to result in disease progression that would require withdrawal of the subject.
7. HIV infection or other immunodeficiency.
8. Previous lung resection or lung reduction surgery within 1-year.
9. Long term oxygen use defined as oxygen therapy prescribed for greater than 12 hours per day.
10. Pulmonary rehabilitation unless such treatment has been stable for at least 4 weeks and remains stable during the study.
11. History of or current malignancy of any organ system, treated or untreated within the past 5 years, except for localized basal or squamous cell carcinoma of the skin.
12. Significant psychiatric disease that would likely result in the subject not being able to complete the study, in the opinion of the Investigator.
13. Findings on physical examination that an investigator considers to be clinically significant.
14. Known alanine aminotransferase (ALT) ≥ 2 × upper limit of normal (ULN), alkaline phosphatase and/or bilirubin > 1.5 × ULN (isolated bilirubin > 1.5 × ULN is acceptable if fractionated bilirubin < 35%).
15. Known diagnosis of severe chronic kidney disease.
16. Any other known abnormal clinical, cardiac or laboratory (hematology, biochemistry or viral) findings, deemed by an investigator to be clinically significantly abnormal.
17. Use of prohibited medications, including nebulized medication, within the time intervals.
18. Current or history of drug or alcohol abuse within the past 5 years.
19. Women who are breast feeding.
20. Use of an experimental drug within 30 days or 5 half-lives, whichever is longer, and/or participation in a study treatment-free follow-up phase of a clinical study within 30 days.
21. Use of an experimental medical device or participation in a follow-up phase of an experimental medical device clinical study within 30 days.
22. Affiliation with the investigator site, including an Investigator, Sub-Investigator, study coordinator, study nurse, other employee of participating investigator or study site or a family member of the aforementioned.
23. A disclosed history or one known to the Investigator of significant noncompliance in previous investigational studies or with prescribed medications.
24. Any other reason that the Investigator considers makes the subject unsuitable to participate.

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2024-06-11 (Actual); Primary Completion 2024-11-26 (Actual); Study Completion 2024-12-03 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Midwest Chest Consultants, Saint Charles, Missouri, United States

IPD SHARING:
Plan to Share IPD: No
There are no plans to make individual participant data available to other researchers.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Following the informed consent process, screening assessments were completed at visits 1 and 2.
Pre-assignment Details: If any inclusion criteria were not met during screening at visit 1 or 2, the subject was not treated with study medication.
  Study medication was dispensed and administered at visit 2 after all eligibility criteria were met.
Groups:
- Ensifentrine 3 mg BID: Inhaled ensifentrine twice daily (BID) for 12 weeks via standard jet nebulizer in addition to standard dual (LAMA/LABA) or triple (LAMA/LABA/ICS) therapy.
  Eligible subjects received ensifentrine.
Period: Overall Study
Arm/Group | Ensifentrine 3 mg BID
Started (Signed the informed consent form and administered treatment at visit 2.) | 20
Completed (Completed 12 weeks of treatment.) | 18
Not Completed | 2
Not completed — Withdrawal by Subject | 2

BASELINE CHARACTERISTICS:
Population: The full analysis set (FAS) included all subjects administered the study medication at visit 2 (day 1), and had a CAT completed at baseline and from at least one post-treatment visit.
Arm/Group | Ensifentrine 3 mg BID
Number analyzed (Participants) | 18
Age, Continuous [Median (Full Range); unit: years] | 73 [57 to 79]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 10
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 18
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 18
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 18
Mean baseline CAT score [Mean (Standard Deviation); unit: units on a scale] — The COPD Assessment Test(tm) (CAT) is a one-page, 8-item questionnaire completed by patients diagnosed with COPD. When completing the questionnaire, individuals rate their experience on a 6-point scale, ranging from 0 (no impairment) to 5 (maximum impairment) with a scoring range of 0-40. Higher scores indicate greater disease impact.
  units on a scale | 18.3 (6.4)

OUTCOME MEASURES:

1. Primary Outcome: The Proportion of CAT Score Responders in the Full Analysis Set at Week 12
Description: Responders are defined as an improvement (decrease) from baseline of ≥2 points. The COPD Assessment Test(tm) (CAT) is a one-page, 8-item questionnaire suitable for completion by patients diagnosed with COPD. When completing the questionnaire, individuals rate their experience on a 6-point scale, ranging from 0 (no impairment) to 5 (maximum impairment) with a scoring range of 0-40. Higher scores indicate greater disease impact. The individual items are: Cough, Mucus, Chest Tight, Breathless, Limited Activities, Confident, Sleep and Energy). CAT was self-completed at baseline, week 6 and week 12.
Time Frame: 12 Weeks
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Ensifentrine 3 mg BID
Number analyzed (Participants) | 18
Participants | 12
Statistical Analysis 1: Comparison: Ensifentrine 3 mg BID; Test type: Other — The proportion of subjects classified as responders at week 12, standard errors, and corresponding 95% CI was estimated by negative binomial regression with background therapy (LABA/LAMA or LABA/LAMA/ICS) included as a fixed effect, and with baseline CAT score included as a covariate. The scale parameter in the negative binomial model was held fixed by specifying a noscale option; Negative binomial regression = 67.0, 95% CI 2-sided [38.0 to 100.0] — A two-sided unadjusted 95% confidence interval for the proportion was used to determine study success with the lower bound of the CI > 0 indicating success

2. Secondary Outcome: The Proportion of CAT Score Responders in the Full Analysis Set at Week 6
Description: Responders are defined as an improvement (decrease) from baseline of ≥2 points. The COPD Assessment Test (CAT) is a one-page, 8-item questionnaire suitable for completion by patients diagnosed with COPD. When completing the questionnaire, individuals rate their experience on a 6-point scale, ranging from 0 (no impairment) to 5 (maximum impairment) with a scoring range of 0-40. Higher scores indicate greater disease impact. The individual items are: Cough, Mucus, Chest Tight, Breathless, Limited Activities, Confident, Sleep and Energy). CAT was self-completed at baseline, week 6 and week 12.
Time Frame: 6 Weeks
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Ensifentrine 3 mg BID
Number analyzed (Participants) | 18
Participants | 8
Statistical Analysis 1: Comparison: Ensifentrine 3 mg BID; Test type: Other — The proportion of subjects classified as responders at week 6, standard errors, and corresponding 95% CI was estimated by negative binomial regression with background therapy (LABA/LAMA or LABA/LAMA/ICS) included as a fixed effect, and with baseline CAT score included as a covariate. The scale parameter in the negative binomial model was held fixed by specifying a noscale option; Negative binomial regression = 44.4, 95% CI 2-sided [22.0 to 89.5] — [estimate comment as in outcome 1, analysis 1]

3. Secondary Outcome: Mean Change From Baseline - CAT Score in the Full Analysis Set
Description: The COPD Assessment Test (CAT) is a one-page, 8-item questionnaire suitable for completion by patients diagnosed with COPD. When completing the questionnaire, individuals rate their experience on a 6-point scale, ranging from 0 (no impairment) to 5 (maximum impairment) with a scoring range of 0-40. Higher scores indicate greater disease impact. The individual items are: Cough, Mucus, Chest Tight, Breathless, Limited Activities, Confident, Sleep and Energy). CAT was self-completed at baseline, week 6 and week 12. A decrease from baseline indicates an improvement in COPD symptoms.
Time Frame: At week 6 and week 12
Population: as for baseline characteristics
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Ensifentrine 3 mg BID
Number analyzed (Participants) | 18
units on a scale
  CAT score at week 6 (mean change from baseline) | -1.5 [-4.0 to 1.1]
  CAT score at week 12 (mean change from baseline) | -2.3 [-4.0 to -0.6]

4. Secondary Outcome: Mean Change From Baseline - CAT Individual Item (1, Cough) in the Full Analysis Set
Description: The COPD Assessment Test (CAT) is a one-page, 8-item questionnaire suitable for completion by patients diagnosed with COPD. When completing the questionnaire, individuals rate their experience on a 6-point scale, ranging from 0 (no impairment) to 5 (maximum impairment) with a scoring range of 0-40. Higher scores indicate greater disease impact.
  Question 1: (0) I never cough → (5) I cough all the time. CAT was self-completed at baseline, week 6 and week 12.
Time Frame: At week 6 and week 12
Population: as for baseline characteristics
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Ensifentrine 3 mg BID
Number analyzed (Participants) | 18
units on a scale
  CAT question 1 (cough) at week 6 (mean change from baseline) | -0.2 [-0.7 to 0.3]
  CAT question 1 (cough) at week 12 (mean change from baseline) | -0.3 [-0.9 to 0.4]

5. Secondary Outcome: Mean Change From Baseline - CAT Individual Item (2, Mucus) in the Full Analysis Set
Description: The COPD Assessment Test (CAT) is a one-page, 8-item questionnaire suitable for completion by patients diagnosed with COPD. When completing the questionnaire, individuals rate their experience on a 6-point scale, ranging from 0 (no impairment) to 5 (maximum impairment) with a scoring range of 0-40. Higher scores indicate greater disease impact.
  Question 2: (0) I have no phlegm (mucus) in my chest at all → (5) My chest is completely full of phlegm (mucus) CAT was self-completed at baseline, week 6 and week 12.
Time Frame: At week 6 and week 12
Population: as for baseline characteristics
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Ensifentrine 3 mg BID
Number analyzed (Participants) | 18
units on a scale
  CAT question 2 (mucus) at week 6 (mean change from baseline) | 0.0 [-0.7 to 0.6]
  CAT question 2 (mucus) at week 12 (mean change from baseline) | -0.5 [-1.1 to 0.0]

6. Other Pre Specified Outcome: Mean Change From Baseline in Blood Pressure in the Safety Analysis Set
Description: Vital signs were assessed at baseline, week 6 and week 12. Week 12 is reported. Determine any clinically significant change from baseline in systolic and diastolic blood pressure.
Time Frame: 12 Weeks
Population: The safety analysis set (SAS) included all subjects who were administered the study medication at day 1 (n=20). However, 2 subjects did not complete week 6 and week 12 visits and did not have a change from baseline calculated.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Ensifentrine 3 mg BID
Number analyzed (Participants) | 18
mmHg
  Systolic blood pressure at week 12 (mean change from baseline) | 1.2 (15.08)
  Diastolic blood pressure at week 12 (mean change from baseline) | 2.8 (10.37)

7. Other Pre Specified Outcome: Mean Change From Baseline in Pulse Rate in the Safety Analysis Set
Description: Vital signs were assessed at baseline, week 6 and week 12. Week 12 is reported. Determine any clinically significant change from baseline in pulse rate.
Time Frame: 12 Weeks
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: bpm
Arm/Group | Ensifentrine 3 mg BID
Number analyzed (Participants) | 18
bpm | 2.9 (11.11)

8. Secondary Outcome: Mean Change From Baseline - CAT Individual Item (3, Chest Tight) in the Full Analysis Set
Description: The COPD Assessment Test (CAT) is a one-page, 8-item questionnaire suitable for completion by patients diagnosed with COPD. When completing the questionnaire, individuals rate their experience on a 6-point scale, ranging from 0 (no impairment) to 5 (maximum impairment) with a scoring range of 0-40. Higher scores indicate greater disease impact.
  Question 3: (0) My chest does not feel tight at all → (5) My chest feels very tight CAT was self-completed at baseline, week 6 and week 12.
Time Frame: At week 6 and week 12
Population: as for baseline characteristics
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Ensifentrine 3 mg BID
Number analyzed (Participants) | 18
units on a scale
  CAT question 3 (chest tight) at week 6 (mean change from baseline) | -0.3 [-0.7 to 0.1]
  CAT question 3 (chest tight) at week 12 (mean change from baseline) | -0.4 [-0.8 to 0.1]

9. Secondary Outcome: Mean Change From Baseline - CAT Individual Item (4, Breathless) in the Full Analysis Set
Description: The COPD Assessment Test (CAT) is a one-page, 8-item questionnaire suitable for completion by patients diagnosed with COPD. When completing the questionnaire, individuals rate their experience on a 6-point scale, ranging from 0 (no impairment) to 5 (maximum impairment) with a scoring range of 0-40. Higher scores indicate greater disease impact.
  Question 4: (0) When I walk up a hill or one flight of stairs I am not breathless → (5) When I walk up a hill or one flight of stairs I am very breathless CAT was self-completed at baseline, week 6 and week 12.
Time Frame: At week 6 and week 12
Population: as for baseline characteristics
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Ensifentrine 3 mg BID
Number analyzed (Participants) | 18
units on a scale
  CAT question 4 (breathless) at week 6 (mean change from baseline) | -0.9 [-1.6 to -0.2]
  CAT question 4 (breathless) at week 12 (mean change from baseline) | -0.5 [-1.0 to 0.0]

10. Secondary Outcome: Mean Change From Baseline - CAT Individual Item (5, Activities) in the Full Analysis Set
Description: The COPD Assessment Test (CAT) is a one-page, 8-item questionnaire suitable for completion by patients diagnosed with COPD. When completing the questionnaire, individuals rate their experience on a 6-point scale, ranging from 0 (no impairment) to 5 (maximum impairment) with a scoring range of 0-40. Higher scores indicate greater disease impact.
  Question 5: (0) I am not limited doing any activities at home → (5) I am very limited doing activities at home CAT was self-completed at baseline, week 6 and week 12.
Time Frame: At week 6 and week 12
Population: as for baseline characteristics
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Ensifentrine 3 mg BID
Number analyzed (Participants) | 18
units on a scale
  CAT question 5 (activities) at week 6 (mean change from baseline) | -0.2 [-0.7 to 0.2]
  CAT question 5 (activities) at week 12 (mean change from baseline) | -0.3 [-0.8 to 0.1]

11. Secondary Outcome: Mean Change From Baseline - CAT Individual Item (6, Confidence) in the Full Analysis Set
Description: The COPD Assessment Test (CAT) is a one-page, 8-item questionnaire suitable for completion by patients diagnosed with COPD. When completing the questionnaire, individuals rate their experience on a 6-point scale, ranging from 0 (no impairment) to 5 (maximum impairment) with a scoring range of 0-40. Higher scores indicate greater disease impact.
  Question 6: (0) I am confident leaving my home despite my lung condition → (5) I am not at all confident leaving my home because of my lung condition CAT was self-completed at baseline, week 6 and week 12.
Time Frame: At week 6 and week 12
Population: as for baseline characteristics
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Ensifentrine 3 mg BID
Number analyzed (Participants) | 18
units on a scale
  CAT question 6 (confidence) at week 6 (mean change from baseline) | 0.1 [-0.5 to 0.8]
  CAT question 6 (confidence) at week 12 (mean change from baseline) | -0.2 [-0.8 to 0.4]

12. Secondary Outcome: Mean Change From Baseline - CAT Individual Item (7, Sleep) in the Full Analysis Set
Description: The COPD Assessment Test (CAT) is a one-page, 8-item questionnaire suitable for completion by patients diagnosed with COPD. When completing the questionnaire, individuals rate their experience on a 6-point scale, ranging from 0 (no impairment) to 5 (maximum impairment) with a scoring range of 0-40. Higher scores indicate greater disease impact.
  Question 7: (0) I sleep soundly → (5) I don't sleep soundly because of my lung condition CAT was self-completed at baseline, week 6 and week 12.
Time Frame: At week 6 and week 12
Population: as for baseline characteristics
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Ensifentrine 3 mg BID
Number analyzed (Participants) | 18
units on a scale
  CAT question 7 (sleep) at week 6 (mean change from baseline) | 0.0 [-0.5 to 0.5]
  CAT question 7 (sleep) at week 12 (mean change from baseline) | 0.2 [-0.2 to 0.5]

13. Secondary Outcome: Mean Change From Baseline - CAT Individual Item (8, Energy) in the Full Analysis Set
Description: The COPD Assessment Test (CAT) is a one-page, 8-item questionnaire suitable for completion by patients diagnosed with COPD. When completing the questionnaire, individuals rate their experience on a 6-point scale, ranging from 0 (no impairment) to 5 (maximum impairment) with a scoring range of 0-40. Higher scores indicate greater disease impact.
  Question 8: (0) I have lots of energy → (5) I have no energy at all CAT was self-completed at baseline, week 6 and week 12.
Time Frame: At week 6 and week 12
Population: as for baseline characteristics
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Ensifentrine 3 mg BID
Number analyzed (Participants) | 18
units on a scale
  CAT question 8 (energy) at week 6 (mean change from baseline) | 0.0 [-0.5 to 0.6]
  CAT question 8 (energy) at week 12 (mean change from baseline) | -0.2 [-0.7 to 0.2]

ADVERSE EVENTS:
Time Frame: 12 weeks
Arm/Group | Ensifentrine 3 mg BID
All-Cause Mortality (participants affected / at risk) | 0/20
Serious Adverse Events (participants affected / at risk) | 0/20
Other Adverse Events (participants affected / at risk) | 0/20

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (2):
  • Study Protocol (2024-08-19): https://cdn.clinicaltrials.gov/large-docs/93/NCT06460493/Prot_000.pdf
  • Statistical Analysis Plan (2024-12-11): https://cdn.clinicaltrials.gov/large-docs/93/NCT06460493/SAP_001.pdf